CLINICAL TRIAL: NCT01759173
Title: Evaluate the Effectiveness of Brain Network Activation (BNA™) Technology in the Management of Sport Related Concussion in the College Age Athletes
Brief Title: Evaluate the Effectiveness of Brain Network Activation (BNA™) Technology in the Management of Sport Related Concussion
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Collaborators: York University (Other)
Responsible Party: Sponsor
Other Study IDs: ELM-18
Record Dates: First submitted 2012-12-03; First posted 2013-01-03 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Minor Traumatic Brain Injury (TBI)
Keywords: Minor traumatic brain injury (TBI); Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- college athletes

SUMMARY:
Currently, there is no direct, reliable, bed-side, and non-invasive method for assessing changes in brain activity associated with concussion. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a noninvasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA™) to temporally and spatially map brain function, connectivity and synchronization.

The proposed study will provide additional evidence for the utility and contribution of the BNA™ test (reflecting temporal and spatial changes in brain activity as well as brain functional connectivity associated with concussion) in concussion management.

ELIGIBILITY:
Inclusion Criteria:

* Age 17-24, both genders, enrolled in a recognized college and members of a sport team of their school.

Exclusion Criteria:

Current or history of any of the following:

* TBI (i.e., Glasgow Coma Scale <13) or brain surgery
* Any psychiatric disorder
* Any Neurological disorder
* Substance abuse
* Special education
* Any medication affecting CNS
* Significant sensory deficits such as deafness or blindness
* Residual symptoms or deficits related to a previous concussion

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 200-300 athletes from 3-9 college sport teams, from both genders, aged 17-24 years.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in BNA™ measures during the sport season in both concussed and non concussed athletes compared to pre season BNA™ baseline measures. | an average of 1 year
Correlation of the BNA measures in both concussed and non concussed athletes to the clinical diagnosis. | an average of 1 year
To assess the clinical utility of changes in BNA in assisting with clinical decision-making. | an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Fallah, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada